CLINICAL TRIAL: NCT02937090
Title: The Cross-sectional Study of Intestinal Microbiota in Women With Polycystic Ovary Syndrome and Its Association With Clinical and Biological Parameters
Brief Title: Intestinal Microbiota Survey of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: PCOS2016
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Intestinal Microbiota
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Polycystic Ovary Syndrome: Premenopausal women between 18-40 years of age.
  Diagnosed with PCOS using Rotterdam criteria (meet 2 of the 3):
  1. chronic oligo- or amenorrhea (irregular periods during more than a year in combination with a cycle length longer than 35 days);
  2. total or free T levels above the reference interval and/or excessive facial hair, acne;
  3. transvaginal ultrasound with polycystic ovaries.
  Exclusion of common medical disorders (normal thyroid function tests and serum prolactin and exclusion of 21-hydroxylase deficiency).
  Interventions: Other: Blood Draw; Other: Stool collection
- Control: Women matched for age and BMI.
  Interventions: Other: Blood Draw; Other: Stool collection

INTERVENTIONS:
Other: Blood Draw — Blood sample will be drawn from participants at study entry.
Other: Stool collection — Stool will be collected from participants at study entry.

SUMMARY:
Polycystic Ovary Syndrome is kind of disease with unclear etiology. Recent studies on intestinal microbiota have raised the possibility that dysbiosis of intestinal microbiota maybe a novel theory for the development of Polycystic Ovary Syndrome. Hence, the investigators will compare the intestinal microbiota composition and diversity in PCOS with age, BMI-matched control and then assess whether intestinal microbiota modification is associated with clinical and biological parameters.

DETAILED DESCRIPTION:
The goal of this study is to investigate and compare the composition of the intestinal microbiota in patients with PCOS and age, BMI-matched control. In addition, the investigators will investigate the relationship between alterations in the intestinal microbiota, clinical phenotype, biochemical analysis, body composition, inflammation and food consumption habit. The investigators hypothesize that alterations in the intestinal microbiota are associated with increased immune activation and progression of PCOS. Based on this hypothesis, the investigators propose the following aims:

Aim 1. Identify and enroll cohort with PCOS and age, BMI-matched control to study the role of intestinal microbiota on the development of PCOS.

1. Enroll participants at Drum Tower Hospital. Identify and classify participants through initial clinical evaluation, collect clinical metadata, obtain and process blood and stool samples for analysis.
2. Characterize the intestinal microbiota through quantitative PCR and high throughput sequencing analysis of stool specimens in participants.

Aim 2. Compare sequencing results and metagenomic analysis for study groups with particular attention to bacterial composition and metabolic capacity associated with energy harvest, lipid and carbohydrate transport, enhancement of epithelial barrier integrity and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal between 18-40 years of age.
2. Exclusion of other etiologies for infertility.

Exclusion Criteria:

1. During the pregnancy and lactation period.
2. Use of antibiotics within 3 months.
3. Regular use of proton pump inhibitors, laxatives or pro-prebiotics.
4. Previous history of gastrointestinal surgery or disease (such as peptic ulcer, irritable bowel syndrome, inflammatory bowel disease or other gastrointestinal disorder).
5. Major changes in eating habits within the past 3 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Polycystic Ovary Syndrome patients and age, BMI-matched women.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiota of stool samples of PCOS and age, BMI-matched control will be identified by quantitative analysis. | an average of 1 month

SECONDARY OUTCOMES:
Correlation of intestinal microbiota composition with biological parameters of PCOS patients will be assessed. | an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No